CLINICAL TRIAL: NCT07236931
Title: Clinical Study of Selinexor-Based Chemotherapy With Minimal or No Cytotoxic Agents in Treatment-Naïve AML Patients Unsuitable for Intensive Therapy: Focusing on Rapid Reduction of Blast Cells
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donghua Zhang (Other)
Responsible Party: Sponsor-Investigator, Donghua Zhang, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZ1962-B
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: AML (Acute Myeloid Leukemia)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): selinexor (X), azacitidine (A), and venetoclax (B) - the XAB regimen
  Interventions: Drug: the XAB regimen

INTERVENTIONS:
Drug: the XAB regimen — the XAB regimen: a chemotherapy-free or low-dose chemotherapy regimen containing selinexor (X), azacitidine (A), and venetoclax (B)

SUMMARY:
This study aims to evaluate the efficacy and safety of selinexor-based chemotherapy-sparing regimens (including chemotherapy-free or dose-reduced approaches) in optimizing therapeutic strategies for treatment-naïve acute myeloid leukemia patients deemed unfit for intensive induction therapy. The investigation will focus on dynamic blast clearance patterns and early toxicity profiles to inform timely treatment adaptation during the critical induction window.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed acute myeloid leukemia (AML) patients Ineligible or unwilling to receive intensive chemotherapy .①Patients deemed ineligible for intensive chemotherapy must meet the following criteria: Age 18 to 74 years with at least one of the following comorbidities; Eastern Cooperative Oncology Group (ECOG) performance status ≥3; Cardiac history requiring treatment for congestive heart failure; Left ventricular ejection fraction ≤50%; Chronic stable angina; Diffusing capacity of the lungs for carbon monoxide (DLCO) ≤65% or forced expiratory volume in 1 second (FEV1) ≤65%; Creatinine clearance ≥30 mL/min to <45 mL/min (Cockcroft-Gault formula); Moderate hepatic impairment: total bilirubin >1.5 to ≤3.0 × upper limit of normal (ULN); ②Other investigator-assessed comorbidities that preclude safe administration of intensive chemotherapy.
2. Hepatic function must meet the following criteria: Aspartate aminotransferase (AST) ≤3.0 × upper limit of normal (ULN); Alanine aminotransferase (ALT) ≤3.0 × ULN; Total bilirubin ≤3.0 × ULN. (unless deemed attributable to leukemic organ involvement)
3. Renal function must meet the following criterion: Creatinine clearance ≥30 mL/min calculated using the Cockcroft-Gault formula.
4. No history of drug allergies within the protocol.
5. Participants with plans for pregnancy must agree to use contraception before enrollment in the study and for six months after the study ends. If a participant becomes pregnant or suspects pregnancy, she must immediately notify the investigator.
6. The participant understands and signs the informed consent form.

Exclusion Criteria:

1. A definitive diagnosis of Acute Promyelocytic Leukemia (APL).
2. Age <18 years or ≥75 years.
3. The participant has previously received any treatment for acute myeloid leukemia (AML), except for hydroxyurea.
4. Uncontrolled active infections (including bacterial, fungal, or viral infections) that are clinically significant and refractory to medical therapy.
5. Currently participating in another clinical study or planning to initiate treatment in this study within less than 4 weeks after the completion of therapy in a prior clinical study.
6. Patients who have other malignancies that require treatment.
7. A history of allergy to the study drugs.
8. Female participants who are pregnant or breastfeeding.
9. Human immunodeficiency virus (HIV) infection or syphilis infection.
10. Active hepatitis that remains uncontrolled despite active antiviral therapy (positive for hepatitis B virus deoxyribonucleic acid [HBV DNA] or hepatitis C virus ribonucleic acid [HCV RNA]).
11. Patients with persistent positivity for Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 (excluding those who have transitioned from positive to negative).
12. Conditions that the investigator considers may increase the risk to participants or interfere with the study results.
13. Other conditions that the investigator deems the participant unsuitable for enrollment in this study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1，3，6，12，18，24 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China